CLINICAL TRIAL: NCT03408197
Title: Comparison of Two Warming Methods in Knee Arthroplasty. A Prospective, Randomized Non-inferiority Trial.
Brief Title: Two Warming Methods in Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R17136
Record Dates: First submitted 2018-01-17; First posted 2018-01-23 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Hypothermia, Accidental
Keywords: inadvertent, intraoperative hypothermia, prewarming; core temperature monitoring
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EasyWarm (Experimental)
  Interventions: Device: EasyWarm
- BairHugger (Active Comparator)
  Interventions: Device: BairHugger

INTERVENTIONS:
Device: EasyWarm — Perioperative warming with EasyWarm to prevent inadvertent hypothermia during anaesthesia
  Arms: EasyWarm
Device: BairHugger — Perioperative warming with BairHugger to prevent inadvertent hypothermia during anaesthesia
  Arms: BairHugger

SUMMARY:
In this study two warming methods will be compared in knee arthroplasty surgery. Barrier EasyWarm will be used in the study group and BairHugger upper body warming blanket in the control group. Both groups will be prewarmed 30 minutes before spinal anaesthesia. In the operating room warming will be continued with the same warming method. Primary end point is core temperature after arriving to post anaesthesia care unit. Hypothesis is that Barrier EasyWarm is not inferior to BairHugger in preventing inadvertent intraoperative hypothermia.

Few methods exist to measure the core temperature non-invasively. Zero-heat-flux technique is used in this study. During the study we will test the accuracy of the 3M BairHugger Temperature Monitoring System by placing two sensors onto the patients (n = 30) fore head. After that the accuracy of the Dräger Tcore is examined by comparing it with the 3M BairHugger Temperature Monitoring System. So the patients (n=30) have both these different core temperature monitoring systems on their foreheads. This observational monitoring study is performed from the patient number 80 until the end.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-40
* ASA class I-III
* elective primary unilateral kneearthroplasty
* spinal anaesthesia

Exclusion Criteria:

* ASA class > III
* unstable coronary artery disease
* revision surgery, bilateral arthroplasty
* general anaesthesia
* decreased mental status

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Core temperature after arriving to the post-anaesthesia care unit | one hour

CONTACTS AND LOCATIONS:
Overall Officials: Maija-Liisa Kalliomäki, Study Director — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lauronen SL, Kalliovalkama J, Aho A, Makinen MT, Huhtala H, Yli-Hankala AM, Kalliomaki ML. Self-warming blanket versus forced-air warming blanket during total knee arthroplasty under spinal anaesthesia: A randomised non-inferiority trial. Acta Anaesthesiol Scand. 2023 Sep;67(8):1102-1109. doi: 10.1111/aas.14283. Epub 2023 May 28. PMID 37246242
- [Derived] Lauronen SL, Kalliomaki ML, Kalliovalkama J, Aho A, Huhtala H, Yli-Hankala AM, Makinen MT. Comparison of zero heat flux and double sensor thermometers during spinal anaesthesia: a prospective observational study. J Clin Monit Comput. 2022 Oct;36(5):1547-1555. doi: 10.1007/s10877-021-00799-6. Epub 2022 Jan 3. PMID 34978656